CLINICAL TRIAL: NCT06845280
Title: Reliability of Respiratory Variability of Maximal Aortic Blood Flow Velocity Obtained by Ultrasonography-doppler in Patients Followed Up with a Diagnosis of Shock in Intensive Care Unit for Evaluating Fluid Responsiveness in Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Uğur Özdemir, Associate Professor, Ankara University
Other Study IDs: 223S949
Record Dates: First submitted 2024-12-27; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Shock
Keywords: Shock; intensive care; transpulmonary thermodilution; echocardiography
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Shock patients: Critically ill shock patients who require at least 0.2mcg/kg/min noradrenaline, or have lactate levels >4 mEq/L and whose clinical tissue perfusion parameters are deteriorating despite adequate treatment for 6 hours (increasing lactate levels, mottling score, decreasing consciousness... ) will be evaluated for eligibility.

SUMMARY:
Original value: Shock is an important cause of mortality in intensive care units (ICU). Determining whether shock patients will benefit from (intravenous) IV fluid therapy is possible by fluid responsiveness parameters/tests. More than half of the patients being monitored for shock in the ICU are not fluid responders. Especially in patients who do not have the desired response despite appropriate shock treatment for the first 6 hours, continuing IV bolus fluid treatments without performing fluid responsiveness tests may cause an increase in mortality due to hypervolemia and organ edema. Today, these tests can be measured with transpulmonary thermodilution (TPTD) devices. Calibration, installation and evaluation of the device requires expert personnel and its use can cause a significant increase in intensive care workload. Instead of this minimal invasive approach, the respiratory variability of maximal aortic blood flow rate (ΔVaortmax), which can be obtained non-invasively with the use of bedside ultrasonography (USG), can be used as a fluid responsiveness parameter. There is no study on the value of this parameter in adult intensive care patients. Revealing the importance of this parameter as a fluid responsiveness parameter may pave the way for ultrasonography devices, which are already in use with other indications, to be used as an important advanced hemodynamic monitoring tool. For this purpose, this prospective observational study was planned.

Method: This study was planned to be conducted on non-pregnant shock patients who are greater than 18 years and who were admitted to Medical ICU of Ankara University Faculty of Medicine, Department of Internal Medicine Division of Intensive Care. It was planned to establish the TPTD system, which is a standard practice in patients whose shock symptoms did not improve and whose lactate level did not decrease despite appropriate fluid, vasopressor and standard intensive care applications for the first 6 hours, and to compare the fluid responsiveness parameters obtained from this TPTD system with the ΔVaortmax obtained by bedside USG. Within the scope of a 6-12 month study period, it is planned to perform advanced hemodynamic monitoring with TPTD in 60 patients and to compare the obtained measurements with ΔVaortmax measurements with bedside USG. In order to carry out the project, a TPTD device and its thermodilution catheters as well as a standard ultrasonography device with an echocardiography system are needed.

Management: Patients who are admitted with shock to our ICU and who develop shock state during their admission will be evaluated for eligibility for the study. A TPTD system will be installed in patients eligible for the study, and a bedside USG will be performed simultaneously and fluid responsiveness and other clinical and hemodynamic data will be recorded. Data will be analyzed to evaluate whether ΔVaortmax, is a good fluid responsiveness parameter for adult shock patients and to determine a cutoff value to assign volume responsive patients.

Widespread effect: With this project, USG/echocardiography devices, which are already commonly used in ICU's for various purposes, will find a new use as advanced hemodynamic monitoring tools to determine fluid responsiveness during shock states, without incurring additional risks to patiens with minimal additional costs. Importantly, this method may reduce the need for some minimally invasive methods such as transpulmonary thermodilution. The results of our project will be disseminated through oral presentations and articles.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Being admitted to medical intensive care unit of Ankara University Faculty of Medicine
* Having a diagnosis of shock
* Deteriorating shock state after the initial 6 hour despite optimal treatment
* Patients or their relatives are required to read, understand and sign the informed consent form for participation in the study.
* Patients who are expected to stay in intensive care for at least 48 hours

Exclusion Criteria:

* The patient has an identified pregnancy or suspected pregnancy.
* Presence of thrombocytopenia that may prevent catheter placement (platelet count less than 50 thousand/mm3 and not being able to be increased)
* Prolongation of prothrombin time that may prevent catheter placement
* Prolongation of activated partial thromboplastin time that may prevent catheter placement
* Failure to provide jugular or subclavian central venous catheterization
* Clinical conditions that prevent the insertion of an arterial thermistor catheter (edema, hematoma, thrombosis, signs of active infection in the area where the catheter will be inserted) and the inability to insert an arterial thermistor catheter
* The patient is receiving CRRT (Continuous renal replacement therapy)/ECMO (Extracorporeal membrane oxygenation)
* Contraindications to passive leg raising test (axial fractures, intra-abdominal hypertension, increased intra-abdominal pressure, lower extremity amputation)
* Presence of conditions preventing bedside USG (chest wall deformity, inability to position the patient appropriately, inadequate image quality, open wound, infection or dressing on the chest wall preventing transthoracic USG)
* Objection of patients' intensivist to enroll the patient (with a documented reason)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Shock patients monitored in intensive care
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Respiratory variability of maximal aortic blood flow | maxiumum 5 days
  To compare respiratory variability of maximal aortic blood flow obtained by transthoracic echocardiography with fluid responsiveness parameters obtained by transpulmonary thermodilution.

SECONDARY OUTCOMES:
Mortality | Mortality event up to first month after the hemodynamic measurements will be monitored.
  To investigate the relationship between fluid responsiveness measurements and mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Medicine Ibn'i Sina Hospital, Ankara, TR, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Ethics committee will be consulted